CLINICAL TRIAL: NCT06552559
Title: Phase 1/2 Study of Selinexor With Dexamethasone, Ifosfamide, Carboplatin, and Etoposide in Patients Who Have Secondary Central Nervous System Involvement With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: Selinexor With ICE Chemotherapy in Secondary Central Nervous System Involving B-cell Non-Hodgkin Lymphoma
Acronym: SIENA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Korean Society of Hematology (Network)
Responsible Party: Principal Investigator, Kim, Seok Jin, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISL2301
Record Dates: First submitted 2024-08-03; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: B-cell Lymphoma Recurrent; B-cell Lymphoma Refractory; CNS Metastases
Keywords: Non-Hodgkin B-cell lymphoma; Secondary CNS involvement; Selinexor; ICE
MeSH Terms: interventions — selinexor; Ifosfamide; Carboplatin; Etoposide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Phase 1/2 study of selinexor in combination with dexamethasone, ifosfamide, carboplatin, etoposide chemotherapy in patients with secondary central nervous system involving relapsed or refractory B-cell non-Hodgkin lymphoma: a single arm, open label, multicentre study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Selinexor plus ICED (Experimental): Phase 1 part of the study:
  Treatment will be repeated every three weeks.
  * Selinexor: DL1 (40mg)/DL2 (60mg)/DL3 (80mg) PO, day 3, 5, 7
  * Ifosfamide 1500 mg/m(2) infused over 2 h on days 1-3
  * Carboplatin (5 AUC) on day 1
  * Etoposide 100 mg/m(2) on days 1-3
  * Dexamethasome 40 mg PO or IV on days 1-4
  Phase 2 part of the study:
  Treatment will be repeated every three weeks.
  * Selinexor: MTD (determined by phase 1 part of the study) PO, day 3, 5, 7
  * Ifosfamide 1500 mg/m(2) infused over 2 h on days 1-3
  * Carboplatin (5 AUC) on day 1
  * Etoposide 100 mg/m(2) on days 1-3
  * Dexamethasome 40 mg PO or IV on days 1-4
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — Combination chemotherapy
  Other Names: Ifosfamide, carboplatin, etoposide, dexamethasone

SUMMARY:
Secondary involvement of the central nervous system (CNS), such as CNS relapse after treatment or progression during treatment, is a rare but deadly occurrence in patients with B-cell non-Hodgkin lymphoma (NHL), particularly in cases of diffuse large B-cell lymphoma (DLBCL) and transformed follicular lymphoma (FL). Despite the grim prognosis associated with secondary CNS involvement, no definitive treatment strategy exists. Selinexor®, an oral, first-in-class, potent selective inhibitor of nuclear export that binds to XPO1, leads to the nuclear retention of tumor suppressor and growth regulator proteins, as well as topoisomerase II enzymes, thereby restoring their functions. Preclinical studies have also shown that selinexor can sensitize cancer cells to topoisomerase inhibitors, alkylating agents, and steroids. Selinexor has been approved by the Food and Drug Administration for relapsed or refractory DLBCL. We hypothesize that selinexor could work synergistically with ifosfamide (an alkylating agent) and etoposide (a topoisomerase II inhibitor) in the ifosfamide, carboplatin, and etoposide (ICE) regimen. High-dose dexamethasone was added to this regimen to enhance the efficacy of ICE as a salvage regimen for secondary CNS involvement, due to its ability to cross the blood-brain barrier.

This phase I/II study aims to evaluate the efficacy and safety of selinexor in combination with ifosfamide, carboplatin, etoposide (ICE), and dexamethasone in patients with relapsed or refractory B-cell non-Hodgkin lymphoma with secondary CNS involvement.

DETAILED DESCRIPTION:
1. Background Secondary central nervous system (CNS) involvement, such as CNS relapse after treatment or progression involving the CNS during treatment, is a rare but deadly occurrence in patients with B-cell non-Hodgkin lymphoma (NHL), particularly in cases of diffuse large B-cell lymphoma (DLBCL) and transformed follicular lymphoma (FL). Despite the grim prognosis associated with secondary CNS involvement, no definitive treatment strategy has been established. Various salvage treatment regimens followed by autologous stem cell transplantation (ASCT) have been attempted, but their effectiveness remains uncertain due to most data coming from retrospective analyses of small case series, with a lack of prospective studies. Since secondary CNS involvement often coincides with systemic disease progression, high-dose methotrexate (MTX)-based regimens may be inadequate for treating systemic disease progression, although they could be effective against CNS tumor cells. Consequently, ICE/D (ifosfamide 1,500 mg/m2/day on days 1-5, carboplatin AUC 5.5 on day 1, etoposide 100 mg/m2 on days 1-5, and dexamethasone 40 mg/day on days 1-4 every 3 weeks) has emerged as another salvage treatment option due to its proven efficacy for both CNS and systemic disease. However, the outcomes of these regimens, including high-dose MTX and/or ICE/D, are still unsatisfactory, with response rates generally below 30-40%. Moreover, most patients who respond to these treatments eventually experience relapse, even after undergoing consolidative ASCT, highlighting the need for improved complete response rates in salvage regimens.

   Exportin 1 (XPO1/CRM1) serves as a nuclear export protein, facilitating the movement of tumor suppressor and growth regulator proteins, such as TP53, p21, p27, FOXO3, and nucleophosmin 1 (NPM1), from the nucleus to the cytoplasm, leading to their deactivation. XPO1 overexpression is common in various malignancies and correlates with poor prognosis. Additionally, XPO1 is responsible for the cytoplasmic transport of topoisomerase II enzymes, and their cytoplasmic presence is linked to drug resistance, as the separation from DNA prevents topoisomerase II inhibitors from triggering cell death.

   Selinexor® is an orally administered, pioneering selective inhibitor of nuclear export, targeting XPO1 to retain tumor suppressor and growth regulator proteins, along with topoisomerase II enzymes, in the nucleus, thus reinstating their activity. Preclinical studies have shown that selinexor can enhance the sensitivity of cancer cells to topoisomerase inhibitors, alkylating agents, and steroids. Selinexor has been approved by the Food and Drug Administration for the treatment of relapsed or refractory DLBCL. We propose that selinexor could enhance the effectiveness of the ifosfamide, carboplatin, and etoposide (ICE) regimen when combined with ifosfamide (an alkylating agent) and etoposide (a topoisomerase II inhibitor), and have included high-dose dexamethasone to potentially increase ICE's efficacy as a salvage therapy for secondary CNS involvement, due to its ability to cross the blood-brain barrier.
2. Study design Phase: I/II Therapeutic Area: Salvage treatment and maintenance for secondary CNS involvement of B-cell NHL Primary Compound: Selinexor Additional compounds (if applicable): Ifosfamide, carboplatin, etoposide, dexamethasone
3. Phase I In the phase 1 study, patients must complete one therapy cycle (3 weeks) at a given dose level before considering escalation to the next level. Escalation is allowed if the initial three patients at a dose level show no dose-limiting toxicities (DLTs) during the first cycle. If one patient experiences DLTs at a dose level of selinexor, three more patients will be added to that level. Escalation to the next selinexor dose level occurs if only one out of six patients experiences DLTs. However, if two out of six patients experience DLTs, the previous dose level is established as the maximum tolerated dose (MTD). If two of the first three patients experience DLTs, the previous dose is deemed the MTD after treating up to six patients at that dose with no more than two experiencing DLTs. If none or only one of the initial three patients, or one out of six patients at a dose level of selinexor, experience DLTs, the dose will be escalated. If the dose level at 60mg/dose of selinexor is to be increased further, 60mg/dose (DL 2) will be considered the MTD, and this dose will be used in the subsequent phase 2 study.

   Phase 1 part of the study:

   Treatment will be repeated every three weeks. - Selinexor: DL1 (40mg)/DL2 (60mg)/DL3 (80mg) PO, day 3, 5, 7 - Ifosfamide 1500 mg/m(2) infused over 2 h on days 1-3 - Carboplatin (5 AUC) on day 1

   - Etoposide 100 mg/m(2) on days 1-3

   - Dexamethasome 40 mg PO or IV on days 1-4
4. Phase 2 Patients with relapsed or refractory DLBCL or FL involving the CNS may be considered for enrollment. Those eligible for transplantation may undergo ASCT following a minimum of two cycles of the study treatment. Patients ineligible for ASCT may be administered up to six cycles of the study treatment. Additionally, maintenance selinexor may be provided irrespective of ASCT eligibility, provided there is no disease progression after completing selinexor-ICED.

   Phase 2 part of the study:

   Treatment will be repeated every three weeks. - Selinexor: MTD (determined by phase 1 part of the study) PO, day 3, 5, 7

   - Ifosfamide 1500 mg/m(2) infused over 2 h on days 1-3
   * Carboplatin (5 AUC) on day 1
   * Etoposide 100 mg/m(2) on days 1-3
   * Dexamethasome 40 mg PO or IV on days 1-4

6) Study endpoints

Primary Endpoint:

Phase 1 part of the study: To determine the maximum tolerated dose (MTD) and recommended phase 2 dose level (RDL) of Selinexor combined with ifosfamide, carboplatin, etoposide and dexamethasone Phase 2 part of the study: Objective response rate - complete and partial response

Secondary Endpoints:

Phase 1 part of the study: Number of participants with dose limiting toxicities Phase 2 part of the study: Duration of response, Progression-free survival, Overall survival, and safety

7) Statistical analysis Phase 1 part of the study: For phase 1, up to 12 patients for 3 levels of Selinexor (3 patients at each level, one cycle) will be recruited on the basis of 3+3 dose escalation design. The aim of this phase 1 study is to evaluate the safety and adverse events, and to reveal minimal efficacy for the next phase 2 clinical trial; thus, the sample size was not determined based on the statistical power.

Phase 2 part of the study: As the primary endpoint of the phase 2 study is objective response rate (ORR) consisting of complete and partial response at the end-of treatment. Although there is limited data about the ORR for relapsed or refractory secondary CNS involving B-cell NHL, the estimated ORR rates were around 20% for those patients. Thus, the sample size calculation for this study is as follows. P1 as 40% (40% being the response proportion that would imply the treatments warrants further investigation) and P0 as 20% (20% being the usual probability of response while using conventional therapy). According to the Simon's Minimax design, we obtained a sample size of 33 (a = 0.05, b = 0.80). If the ORR is ≤ 4/18, the trial would be stopped. If the ORR is > 4/18, the recruitment of subjects would be continued until the number of 33. Considering 10% drop-out rate, a total of 37 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed B-cell NHL with CNS involvement DLBCL including ABC, GCB or PMBCL subtypes Indolent lymphomas transformed to aggressive lymphomas Follicular lymphomas
* Patients must have received at least one cycles of anthracycline based chemotherapy administered with curative intent
* Patients must be age ≥18 years.
* Patients must have at least one site of measurable disease, 1.5 cm in diameter or greater.
* Patients must have ECOG performance status of 0-2.
* Patients must have laboratory test results within these ranges: Absolute neutrophil count ≥ 1500/mm³, Platelet count ≥ 100,000/mm³, Serum creatinine clearance ≥40 mL/min, Total bilirubin ≤ 1.5x ULN (Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis.), AST (SGOT) and ALT (SGPT) ≤ 2x ULN
* Women of childbearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test prior to selinexor treatment. Male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential.
* Patients must be able to understand and willing to sign a written informed consent document.
* Patients must be able to adhere to the study visit schedule and other protocol requirements.
* Patients must not have any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Patients must not have any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Patients with hepatitis B virus including HBsAg-positive carrier or IgG anti- HBc-positive can be enrolled if they can receive anti-viral prophylaxis

Exclusion Criteria:

* Patients cannot fulfill the above-mentioned inclusion criteria
* Patients with primary CNS lymphoma
* Patients with a prior history with selinexor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of elinexor in phase 1 | Up to 1 year
  Maximum tolerated dose and recommended phase 2 dose level of Selinexor combined with ifosfamide, carboplatin, etoposide and dexamethasone
Objective response rate | Up to 2 years
  Complete and partial response out of participants in phase 2

SECONDARY OUTCOMES:
Duration of response | Uo to 3 years
  Time between the first determined response and the data of porgression

CONTACTS AND LOCATIONS:
Overall Officials: Seok Jin Kim, Study Chair — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Samsung Cancer Research Institute, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No